CLINICAL TRIAL: NCT01579799
Title: The Effect of L-lysine on Human Gastrointestinal Secretion: A Dose-finding Study Applying Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: KEK-ZH-NR. 2012-0005
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Lysine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Dose 0.5 (Active Comparator)
  Interventions: Drug: L-lysine
- Dose 7.5 (Active Comparator)
  Interventions: Drug: L-lysine
- Dose 3 (Active Comparator)
  Interventions: Drug: L-lysine
- Dose 1.2 (Active Comparator)
  Interventions: Drug: L-lysine

INTERVENTIONS:
Drug: L-lysine — Dose finding study for L-lysine

SUMMARY:
This is a pilot dose-finding study, which is performed with a randomized, double-blind, 3-armed, unbalanced, cross-over study design. Three of four different doses of L-lysine Monohydrate (A = 0.5 g, B = 1.2 g, C = 3.0 g and D = 7.5 g) will be applied in a randomized sequence on three different study days in six healthy volunteers. Each study day involves the repeated measurement of gastric content volume, gastric secretion volume and intestinal fluid volume using MRI before and after intragastric infusion of L-lysine Monohydrate test meals. Additionally, symptoms for hunger, fullness, nausea, bloating, abdominal cramps and urge to defecate will be recorded using a scale from 0-10. In parallel, samples of gastric juice to measure intragastric pH and pepsin concentration, samples of venous blood to assess blood pH and haematocrit as well as L-lysine, Serotonin, chloride bicarbonate and albumin plasma concentration and samples of arterialized blood from ear lobe to measure glucose blood concentration will be collected

ELIGIBILITY:
Inclusion criteria: > 18, < 50 years Healthy BMI > 19, <24

Exclusion criteria: Age under 18 or above 50

* Pathologic underweight or overweight (BMI <19 or >24 (kg/m2))
* Previous gastrointestinal, cardio-respiratory (incl. arterial hypertension), hematologic (anaemia), renal, hepatic, atopic, alimentary disease, psychiatric disease, epilepsy, panic attacks, diabetes drug or alcohol abuse, lysinuria, galactosaemia
* Subjects unable to stop medication that alters gut function for 1 week prior to the study, including anticholinergics, calcium canal inhibitors, beta blocker, prokinetics, proton-pump inhibitors, DDV-IV-Inhibitors, Incretin-mimetics, non-steroidal anti-inflammatory drugs, Macrolidantibiotica
* Subjects unable to stop medication within 48 prior the study begins that alters serotonin blood profiles , including paracetamol, cumarine, mephenesin, phenobarbital, acetanilide, ephedrine, amphetamine, phentolamin, phenacetin, methocarbamol, acetylsalicylic acid, levodopa, promethazine, isoniazid, methenamine, streptozocin, chlorpromazine
* Positive helicobacter pylori test
* Previous history of gastrointestinal disease or surgery (excludes appendectomy, hernia repair and anorectal disorders)
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female patients of child bearing age will receive a pregnancy test prior to study)
* Involvement in any other clinical trial during the course of this trial, nor within a period of 14 days prior to its beginning or 14 days after its completion
* Mental capacity (DSM IV, inter alia Claustrophobia), which limits the capability to fulfill the demands of the study
* Known allergy or intolerance against capsaicin, locus bean gum, L-lysine, DOTAREM®, Fructose, Gluten, Galactose Known allergic reaction after prior injection of lidocaine (e.g. at the dentist )
* Known allergic reaction toward methylparaben (E218)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Gastric half-emptying time | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schwizer, Prof. MD, Principal Investigator — University Hospital Zurich, Gastroenterology & Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology, Zurich, Canton of Zurich, Switzerland